CLINICAL TRIAL: NCT00054821
Title: Pathogenesis-Prevention of Post-Traumatic Osteoarthritis (OA): Effects of Distraction and Motion on OA
Brief Title: Prevention of Post-Traumatic Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ned Amendola (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Ned Amendola, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P50AR048939 (NIH); P50AR048939 (NIH); NIAMS-082
Record Dates: First submitted 2003-02-11; First posted 2003-02-13 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Ankle; Ankle Distraction
MeSH Terms: conditions — Osteoarthritis | interventions — Motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A participants will be treated with mechanical distraction with motion
  Interventions: Procedure: Ankle distraction permitting motion
- Group B (Active Comparator): Group B participants will be treated with mechanical distraction without motion
  Interventions: Procedure: Ankle distraction without motion

INTERVENTIONS:
Procedure: Ankle distraction permitting motion — External fixator is applied to ankle joint for 85 - 95 days; ankle motion is permitted
  Arms: Group A
Procedure: Ankle distraction without motion — External fixator is applied to ankel joint for 85 - 95 days; ankle motion is not permitted
  Arms: Group B

SUMMARY:
Joint injury and trauma dramatically increase the risk of developing osteoarthritis (OA). The purpose of this study is to determine what factors lead to decreased pain, improved joint function, and repair of the joint surface in post-traumatic OA.

Study hypotheses: 1) Ankle motion during distraction will result in clinically significant improvements in Ankle Osteoarthritis Scale scores, SF-36 scores, and improved cartilage thickness distribution over the habitually most heavily loaded portion of the articular surface, as compared to the use of distraction without ankle motion. 2a) Ankles with low geometric surface irregularity and greater range of motion will have better preservation of neo-chondroid tissue (increased normalized cartilage thickness and reduced longitudinal compressive strain in the habitually heavily regions of the articular surface) than those with high surface irregularity. 2b) Low geometric surface irregularity and greater range of motion will have reduced habitual focal or regional contact stress elevation. 3) Joints that have better improvements in Ankle Osteoarthritis Scale scores and improved cartilage thickness distribution over habitually heavily loaded portion of the articular surface will have improved normalization of synovial fluid markers of biosynthetic/degradative activity and oxidative stress.

DETAILED DESCRIPTION:
Little work has been done on the pathogenesis and prevention of post-traumatic OA. The human ankle joint provides a unique opportunity for the study of post-traumatic OA because of the low risk of primary OA and the relatively high risk of post-traumatic OA. This study involves a multidisciplinary approach utilizing both laboratory and clinical research to improve understanding of OA and to develop innovative approaches for preventing and treating this disease. Mechanical distraction involves operative placement of specialized pins and rods to hold the joint in place. Some distraction allows for limited motion of the joint, while other distraction holds the joint immobile. The purpose of this study is to elucidate the mechanical factors that lead to restoration of a cartilaginous articular surface, decreased pain, and improved joint function after mechanical distraction of osteoarthritic joints.

Participants in this study will be randomly assigned to one of two treatment groups. Group A will be treated with mechanical distraction with motion; Group B will be treated with mechanical distraction without motion. Participants will be followed for 28 months and will have 11 study visits. Most of the study visits will occur during the first half of the study. State-of-the-art techniques for clinical assessment, articular surface imaging, biomechanical modeling, and biochemical testing will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic isolated ankle OA (unilateral Kellgren grade 3, 4, or 5)
* Skeletally mature (children included if they have no open growth plates)
* Failure of less than 1 year nonoperative treatment, including 3 months of continuous treatment with nonsteroidal anti-inflammatory agents and 3 months of unloading treatment (i.e., unloading brace, crutches, cane, walker)

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2002-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Ankle Osteoarthritis Scale scores | Two years
CT data to measure cartilage distribution over the articular surface and synovial fluid markers of biosynthetic/degradative activity and oxidative stress in response to treatment and comparison to clinical and radiographic changes | Two years
Improved joint function | Two Years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Buckwalter, MD, Principal Investigator — University of Iowa; Thomas D. Brown, PhD, Principal Investigator — University of Iowa
Locations (1):
- Department of Orthopedics and Rehabilitation, University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Buckwalter JA. Sports, joint injury, and posttraumatic osteoarthritis. J Orthop Sports Phys Ther. 2003 Oct;33(10):578-88. doi: 10.2519/jospt.2003.33.10.578. PMID 14620787
- [Background] Buckwalter JA, Brown TD. Joint injury, repair, and remodeling: roles in post-traumatic osteoarthritis. Clin Orthop Relat Res. 2004 Jun;(423):7-16. PMID 15232420